CLINICAL TRIAL: NCT04686903
Title: Prospective Comparison Between Epiduroscopy Procedure, Racz Catheter Procedure and Caudal Epidural Block in Patients With FBSS
Brief Title: EuroPainClinicsStudy IX
Acronym: EPCS IX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Europainclinics z.ú. (Other)
Collaborators: Brno University Hospital (Other); Slovak Academy of Sciences (Other Government); Pavol Jozef Safarik University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03595/2020/OZ-30
Record Dates: First submitted 2020-12-15; First posted 2020-12-29 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Failed Back Surgery Syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome

STUDY DESIGN:
Intervention Model Description: 3 paralel groups: Group A Epiduroscopy in patients with FBSS (50 patients) Group B Racz catheter epidural procedure in patients with FBSS (50 patients) Group C Caudal epidural block in patients with FBSS (50 patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Epiduroscopy (Experimental): Epiduroscopy in patients with FBSS
  Interventions: Procedure: Epiduroscopy treatment
- Racz catheter epidural procedure (Experimental): Racz catheter epidural procedure in patients with FBSS
  Interventions: Procedure: Racz catheter epidural procedure
- Caudal epidural block (Experimental): Caudal epidural block treatment of FBSS
  Interventions: Procedure: Caudal epidural block

INTERVENTIONS:
Procedure: Epiduroscopy treatment — Device Epiduroscop, procedure mecahnical lysis, laser, radiofrequency + drug administration into the epidural space (corticosteroid methylprednisolone acetate 80mg and solution of hyaluronidase 150 I.U. in 10mL of saline) Follow-up: before procedure, 6 months and 12 months after procedure
  Arms: Epiduroscopy
Procedure: Racz catheter epidural procedure — Device Racz catheter, two procedures during clinical trial observation
  * First procedure after enrolment into the study mechanical lysis and drug administration into the epidural space (corticosteroid methylprednisolone acetate 80mg and solution of hyaluronidase 150 I.U. in 10mL of saline)
  * Second procedure after 6 months mechanical lysis + drug administration into the epidural space (corticosteroid methylprednisolone acetate 80mg and solution of hyaluronidase 150 I.U. in 10mL of saline)
  Arms: Racz catheter epidural procedure
Procedure: Caudal epidural block — Technique Caudal epidural block
  Three procedures during clinical trial observation :
  * First procedure after enrolment into the study drug administration into the epidural space (corticosteroid methylprednisolone acetate 80mg and solution of hyaluronidase 150 I.U. in 10mL of saline)
  * Second procedure after 4 months drug administration into the epidural space (corticosteroid methylprednisolone acetate 80mg)
  * Third procedure after 8 months drug administration into the epidural space (corticosteroid methylprednisolone acetate 80mg)
  Arms: Caudal epidural block

SUMMARY:
Prospective comparison between epiduroscopy procedure, Racz catheter procedure and caudal epidural block in patients with FBSS

DETAILED DESCRIPTION:
I. Epiduroscopy is an advanced proven diagnostic and therapeutic method for chronic radicular pain after spinal surgery. Moreover, this method is frequently used in patients with chronic low back pain conditions without previous spine surgery also known as "virgin back". Epiduroscopy allows by optical fiber technology and skiascopy imaging the exact examination of the epidural space and subsequently mechanical lysis (with advanced interventional options by laser, radiofrequency, balloon techniques etc.) and/or drug administration to the target point.

II. The Racz catheter procedure is based on epidural neurolysis. It is used to release some of the adhesions or scar tissue which surround entrapped nerves in the epidural space of the spine. This state could be caused by chronic inflammatory adhesions or by healing mechanisms after spine surgery - scars. Mechanical liberation of epidural space further allows better administration and targeting of drugs as corticoids or hyaluronidase. This technique is performed under fluoroscopy imaging. Suitable epidurogram and skiascopy confirm appropriate catheter position during procedure.

III. The caudal epidural block involves placing a needle through the sacral hiatus to deliver medications into the epidural space. This approach to the epidural space is popular in managing a wide variety of chronic pain conditions in adults, especially chronic low back pain syndromes. Fluoroscopy is considered as a gold standard of needle guidance during procedures in which caudal epidural injections are performed.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 20 and 80
* patients with FBSS (at least 1 - up to 2 lumbar laminectomies) who has radiating pain (VAS >=5) on lower extremities
* those who (only if a signature was obtainable), or whose legal guardian, fully understood the clinical trial details and signed the informed consent form

Exclusion Criteria:

* more than 2 lumbar laminectomies
* patients without previous spine surgery
* patients with a history of other spinal diseases (compression fracture, spondylitis, tumor)
* women with a positive pregnancy test before the trial or who planned to become pregnant within the following 3 years
* other patients viewed as inappropriate by the staff
* disagreement with participation in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline EuroQoL-5 dimension (EQ-5D) value 6m | 6 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change from baseline EuroQoL-5 dimension (EQ-5D) value 12m | 12 months follow-up
  EQ-5D-5L self-care, usual activities, pain/discomfort and anxiety/depression
Change from baseline Visual Analog Pain Scale (VAS) of back pain 6m | 6 months follow-up
  VAS 10 point measurement
Change from baseline Visual Analog Pain Scale (VAS) of back pain 12 m | 12 months follow-up
  VAS 10 point measurement
Oswestry disability index (ODI) 6m | 6 months follow-up
  he ODI self-administered questionnaire measuring 0-100 scale function.'' The questionnaire comprises 10 items, each with 6 levels of response. Each item is scored from 0 to 5, and the total summation is converted to a 0-100 scale. The ODI scores range from 0 to 100, with higher scores indicating severe symptoms.
Oswestry disability index (ODI) 12m | 12 months follow-up
  he ODI self-administered questionnaire measuring 0-100 scale function.'' The questionnaire comprises 10 items, each with 6 levels of response. Each item is scored from 0 to 5, and the total summation is converted to a 0-100 scale. The ODI scores range from 0 to 100, with higher scores indicating severe symptoms.

SECONDARY OUTCOMES:
Before procedure drug usage | before procedure
  drug usage
Postprocedural drug usage | before procedure
  drug usage
Radiation exposure | 12 months follow-up
  Dose of radiation exposure

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Burianek, MD MBA, Study Chair — Europainclinics z.ú.
Locations (1):
- EuroPainClinics, Bardejov, Slovakia

IPD SHARING:
Plan to Share IPD: No
encrypted database